CLINICAL TRIAL: NCT01382277
Title: Rosuvastatin Effect on Reducing Coronary Atherosclerosis Plaques Volume Evaluated by Multi-slice Spiral CT in Patients With Stable Coronary Heart Disease and Hyperlipidemia
Brief Title: Rosuvastatin Effect on Reducing Coronary Atherosclerosis Plaques Volume
Acronym: REDUCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Yong Huo, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REDUCT
Record Dates: First submitted 2011-06-20; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-02

CONDITIONS: Hyperlipidemia; Coronary Artery Disease
MeSH Terms: conditions — Hyperlipidemias; Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rosuvastatin 20 mg (Experimental): Rosuvastatin 20 mg for 76 weeks.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20 mg per day for 76 weeks
  Other Names: Crestor

SUMMARY:
This multicentre, open-label, single-arm Study is to evaluate the effect of Rosuvastatin 20 mg 76 weeks on coronary atherosclerosis plaque versus baseline in Chinese coronary heart disease (CHD) patients with hyperlipidemia by measuring the plaque volume using a 64 slice spiral CT. Effect on blood lipids, hsCRP and Carotid intima-media thickness (CIMT) is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Men or women, aged 18 -75
* Diagnosed with coronary heart disease (CHD) stable angina for more than 1 month and meet the following any one:

  1. History of myocardial infarction.
  2. CHD confirmed by coronary angiography.
  3. Excercise ECG positive for CHD or perfusion defect
  4. One or more main branch of coronary artery stenosis ≥ 50% confirmed by CT scanning.
* Hyperlipidemia (lipid-lowering treatment naïve: LDL-C ≥130mg/dl, or having received lipid-lowering treatment: LDL-C ≥100mg/dl)
* The 64 slice CT shows at least one significant coronary artery stenosis ≥20% with the narrowest ≤60% and meeting the following criteria:

  1. Diameter of coronary artery lesion ≥2mm, length ≥5mm; distance between multiple lesions >1cm
  2. Plaque density <100HU, no calcification
  3. Vascular stenosis (20～60%) caused by plaques
  4. Plaque thickness >1mm
  5. Plaque not in the coronary artery with previous PCI treatment.

Exclusion Criteria:

* Acute myocardial infarction within 6 months
* PCI or CABG therapy within 6 months
* Anticipated PCI or CABG therapy in the following 3 months.
* Tropnin I/Tropnin T higher than ULN
* Cardiac failure NYHA III or above
* Coronary artery left main stenosis >50%
* Emergency coronary angiography(CAG) is needed
* Serious arrhythmia or tachycardia
* Secondary hyperlipidemia
* Familial hypercholestrolemia
* Uncontrolled severe hypertension (≥200/110 mmHg)
* Uncontrolled diabetes (HbA1c ≥9.5%)
* Triglyceride ≥500 mg/dL (5.65 mmol/L)
* Active hepatic disease or hepatic function impairment, ALT≥3ULN
* Serum creatinine >177 µmol/L (2.0 mg/dL)
* Myalgia or blood CK ≥5ULN
* WBC < 4×10e9/L，or PLT < 100*10e9/L。
* Participation in the the course of plan and/or procedure of this study
* Previous participation in the study treatment
* Participation in other clinical studies in the past 3 months
* Pregnant or breast-feeding women, women with child-bearing potential who did not use drugs or devices for contraception, or women with positive urine pregnancy test (human chorionic gonadotropin [HCG])
* History of malignant tumors (exception: recovered more than 10 years or only basal cell carcinoma or squamous cell carcinoma); females with a history of cervical atypical hyperplasia (exception: 3 consecutive cervical smear tests normal prior to enrolment)
* History of alcohol and/or drug abuse in recent 5 years
* Any serious or unstable physical or psychological conditions, in the opinion of the investigator, would compromise the safety of the patient or the participation in this study
* Use of concomitant medications prohibited in this study ( Erythromycin, clarithromycin, erythromycin ethylsuccinate, sulfaphenazole; Fluconazole, ketoconazole, itraconazole; Niacin / nicotinic acid(including vitamins/food additives containing niacin / nicotinic acid >50mg), probucol, clofibrate, cholestyramine, colestipol hydrochloride, ezetimibe, fenofibrate, gemfibrozil, atorvastatin(exception: study medication)，lovastatin, pravastatin, rosuvastatin (exception: study medication) , Simvastatin, fluvastatin, fish oil (any dose), lipid-lowering supplements and food additives; Cyclosporine; Protease inhibitors)
* Use of periodic hormone replacement treatment(HRT), oral contraceptives(OCTs), long-acting progesterone, or in recent 3 months non-periodic HRT or OCTs
* Patients with any condition which, in the investigator's judgment, might increase the risk to the subject for any adverse event or abnormal laboratory finding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in coronary atherosclerosis plaque volume using a 64 slice spiral CT at 76 weeks | 76 weeks

SECONDARY OUTCOMES:
Change from baseline in blood lipids at 26 weeks | 26 weeks
Change from baseline in hsCRP at 26 weeks | 26 weeks
Change from baseline in Carotid intima-media thickness at 76 weeks | 76 weeks
Number of participants with adverse events and abnormal laboratory safety markers. | 76 weeks
Change from baseline in blood lipids at 52 weeks | 52 weeks
Change from baseline in blood lipids at 76 weeks | 76 weeks
Change from baseline in hsCRP at 52 weeks | 52 weeks
Change from baseline in hsCRP at 76 weeks | 76 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Division of Cardiology, Peking University First Hospital, Beijing